CLINICAL TRIAL: NCT00801554
Title: A Characterization Study of Individuals With Autism Spectrum Disorders
Brief Title: Autism Spectrum Disorders (ASD) Characterization Study
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD; Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2007-P-001951
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorder; ASD; Autism; Asperger's Syndrome; PDD-NOS; Pervasive Developmental Disorders- Not Otherwise Specified; Adults; Children
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ASD: Children and adults with Autism Spectrum Disorders.
- Non-ASD: Healthy volunteers who have never been diagnosed with an Autism Spectrum Disorder in their lifetime.

SUMMARY:
The overarching aim of the study is to characterize children and adults with ASDs, and compare them with age-matched controls in relation to their functioning in family, academic, employment, and social spheres. Subjects will be comprehensively assessed in multiple non-overlapping domains of functioning, using psychiatric, cognitive, and psychosocial instruments.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-60 years old
* For subjects who have ASD: Meet DSM-IV PDD criteria based on clinical assessment including PDD module of structured interview
* For subjects who have ASD: One parent/guardian available for interviews about each subject. If a parent or guardian is not available, a reliable adult reporter identified by the subject available for an interview
* Full-scale IQ of above 80

Exclusion Criteria:

* Major sensorimotor handicaps (e.g. deafness, blindness)
* Any severely unstable psychiatric conditions including the following: psychosis, suicidality, bipolar disorder, substance use disorders (alcohol or drugs) that would require in-patient hospitalization.
* Inadequate command of the English language.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adults with ASDs.
  Controls: healthy volunteers who have never been diagnosed with an Autism Spectrum Disorder.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Overall level of functioning of children and adults with autism spectrum disorders (ASD) compared to individuals without ASD. | single time point

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States